CLINICAL TRIAL: NCT03444363
Title: Evaluation of Long-Term Effects of Diode Laser Application on Periodontal Healing, Serum C-Reactive Protein and HbA1c Levels in Periodontal Treatment of Uncontrolled Type-2 Diabetic Subjects With Chronic Periodontitis
Brief Title: Periodontal Treatment With Diode Laser in the Patients With Diabetes Melitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Abubekir Eltas, Director, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/104
Record Dates: First submitted 2018-02-15; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus; Periodontal Disease
Keywords: laser; periodontal treatment; systemic inflammation; glycemic control
MeSH Terms: conditions — Diabetes Mellitus; Periodontal Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, controlled.
Who Masked: Participant, Investigator
Masking Description: The results of the study were evaluated in a blinded manner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): SRP plus diode laser (810 nm wavelength, 1 W power)
  Interventions: Device: Laser group
- Control group (Active Comparator): SRP plus placebo
  Interventions: Device: Control group

INTERVENTIONS:
Device: Laser group — Laser application in addition to SRP
  Other Names: Gigaa Laser
  Arms: Study group
Device: Control group — Placebo laser application in addition to SRP
  Arms: Control group

SUMMARY:
This study aimed to investigate the effects of diode laser (DL) in addition to non-surgical periodontal treatment on periodontal parameters, systemic inflammatory response, and serum hemoglobin A1c (HbA1c) level in patients with uncontrolled type 2 diabetes mellitus (T2DM) and chronic periodontitis.

DETAILED DESCRIPTION:
This study was designed as a randomized, controlled, full-mouth, 6-month clinical trial. 37 patients (20 women and 17 men) with uncontrolled T2DM and chronic periodontitis who were selected from among those admitting to Dentistry Faculty of Inonu University and Turgut Ozal Medical Center completed this study. The patients were divided into two groups. The individuals in the control group underwent placebo laser treatment in addition to scaling and root planing (SRP). The individuals in the study group underwent DL (1 W power) in addition to SRP. Clinical index measurements were performed before treatment (T0), 3 months after treatment (T1), and 6 months after treatment (T2). Plaque index (PI), gingival index (GI), bleeding on probing (BOP), clinical attachment level (CAL), and probing depth (PD) were measured to determine periodontal status. HbA1c and C-reactive protein (CRP) levels were also analyzed using blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of type-2 DM according to the ADA criteria for at least two years before the study, HbA1c⩾7%,28
* Having no change in antidiabetic drugs in the last 3 months,
* Having no major diabetes complications (because chronic complications of diabetes complicate metabolic control),
* Presence of generalized CP,29
* Presence of an area with a pocket depth of 4-7 mm in at least four teeth in the upper jaw,
* Presence of at least 20 teeth in the mouth,
* Having no any systemic illness except for DM,
* Having no smoke,
* Receiving no periodontal treatment in the last 12 months,
* Receiving no antibiotics or anti-inflammatory drugs for a long period in the last 6 months,
* Not being pregnant or not to breastfeed,
* Having no third molars.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2014-02-15 (Actual); Study Completion 2014-12-23 (Actual)

PRIMARY OUTCOMES:
Laboratory findings | Six months
  Serum HbA1c levels were measured using the high-performance liquid chromatography method.

SECONDARY OUTCOMES:
Clinical findings | Six months
  Probing depth (PD) was measured the distance between the gingival margin and the deepest aspect of the pocket (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa O Uslu, Dr., Study Chair — Inonu University
Locations (1):
- Abubekir Eltas, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No